CLINICAL TRIAL: NCT01747759
Title: Evaluation of a Preoperative Education in Total Knee Arthroplasty
Acronym: EPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHU-0133
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Knee Osteoarthritis (Knee OA)
Keywords: • Knee osteoarthritis; Total knee arthroplasty; Selfcare; Booklet; Rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Kruskal-Wallis and qualitative parameters (Other): The evaluations will take place at baseline, the day before surgery and 6 weeks post-surgery on knowledge and beliefs scores at each visit and on a satisfaction score on the last one. Quantitative data will be compared between groups by the Kruskal-Wallis and qualitative parameters via Fisher exact test
  Interventions: Other: Kruskal-Wallis and qualitative parameters
- Fisher exact test (Other): The evaluations will take place at baseline, the day before surgery and 6 weeks post-surgery on knowledge and beliefs scores at each visit and on a satisfaction score on the last one. Quantitative data will be compared between groups by the Kruskal-Wallis and qualitative parameters via Fisher exact test
  Interventions: Other: Kruskal-Wallis and qualitative parameters

INTERVENTIONS:
Other: Kruskal-Wallis and qualitative parameters

SUMMARY:
The benefit of preoperative rehabilitation treatment combining physiotherapy and targeted education for patient undergoing Total Knee replacement (TKR) is now well known. Thus, there is lack of validated booklet containing evidence based informations.

Our aim is to assess the impact of an evidence based education pre-operative booklet on patient's knowledge and beliefs. The secondary objectives are to assess the impact of the booklet on patient's satisfaction on the information received, the length of stay in orthopedic surgery and the transfer rate to rehabilitation wards.

To show a difference of 2 points on the knowledge score (range 0-10) between the two groups, with a = 0.05 and a power of 90%, we considered that 44 patients are needed. The evaluations will take place at baseline, the day before surgery and 6 weeks post-surgery on knowledge and beliefs scores at each visit and on a satisfaction score on the last one. Quantitative data will be compared between groups by the Kruskal-Wallis and qualitative parameters via Fisher exact test.

The study protocol was approved by the local Ethic Committee.

DETAILED DESCRIPTION:
The benefit of preoperative rehabilitation treatment combining physiotherapy and targeted education for patient undergoing Total Knee replacement (TKR) is now well known. Thus, there is lack of validated booklet containing evidence based informations.

Our aim is to assess the impact of an evidence based education pre-operative booklet on patient's knowledge and beliefs. The secondary objectives are to assess the impact of the booklet on patient's satisfaction on the information received, the length of stay in orthopedic surgery and the transfer rate to rehabilitation wards.

To show a difference of 2 points on the knowledge score (range 0-10) between the two groups, with a = 0.05 and a power of 90%, we considered that 44 patients are needed. The evaluations will take place at baseline, the day before surgery and 6 weeks post-surgery on knowledge and beliefs scores at each visit and on a satisfaction score on the last one. Quantitative data will be compared between groups by the Kruskal-Wallis and qualitative parameters via Fisher exact test.

The study protocol was approved by the local Ethic Committee.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 55 to 75 Planned total knee arthroplasty

Exclusion Criteria:

* Age under 55 or above 75 Patients institutionalized Patients who have received a total knee arthroplasty of the ipsilateral knee Patient not affiliated to a social security scheme (beneficiary or assignee) Patients with chronic inflammatory rheumatism Cognitive and behavioral issues Disorders of understanding and expression of the French language TKR on complex knee

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
knowledge score | at day 1

SECONDARY OUTCOMES:
pain | Baseline
Primary disability | Baseline
Duration of hospitalization surgery | at day 1
Transfer rate in acute care and rehabilitation, and length of stay | at week 6
Patient's overall satisfaction towards the information received | at week 6
Patient's confidence in its own ability to achieve rehabilitation | at day-1
Patient's knowledge and beliefs about his condition | Baseline, at day-1 and week 6

CONTACTS AND LOCATIONS:
Overall Officials: Stephane DESCAMPS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Eschalier B, Descamps S, Pereira B, Vaillant-Roussel H, Girard G, Boisgard S, Coudeyre E. Randomized blinded trial of standardized written patient information before total knee arthroplasty. PLoS One. 2017 Jul 5;12(7):e0178358. doi: 10.1371/journal.pone.0178358. eCollection 2017. PMID 28678854